CLINICAL TRIAL: NCT01137578
Title: Pilot Study for Assessing Diagnostic Techniques for Central Venous Catheter-related Venous Thromboembolism
Brief Title: Pediatric Catheter-related Thrombosis Imaging Study
Acronym: AESOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CV185-077; 2009-016906-18 (EudraCT Number)
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-11

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — High-Energy Shock Waves; Magnetic Resonance Spectroscopy; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A: US, MRI with contrast, MRI without contrast (Other): Subjects with a central venous catheter (CVC) in place and asymptomatic for a CVC-related DVT to have an Ultrasound (US), Magnetic Resonance Imaging (MRI) with contrast and MRI without contrast performed.
  Interventions: Procedure: Ultrasound; Drug: Magnetic Resonance Imaging with Contrast; Procedure: Magnetic Resonance Imaging without Contrast
- Cohort B: US, MRI with contrast, MRI without contrast (Other): Subjects with a CVC in place either symptomatic for a CVC-related DVT or having an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons to have an Ultrasound, Magnetic Resonance Imaging (MRI) with contrast and MRI without contrast performed.
  Interventions: Procedure: Ultrasound; Drug: Magnetic Resonance Imaging with Contrast; Procedure: Magnetic Resonance Imaging without Contrast
- Cohort C: US, MRI with contrast, MRI without contrast (Other): Subjects with a CVC in place having an MRI for clinical reasons to have an Ultrasound, Magnetic Resonance Imaging (MRI) with contrast and MRI without contrast performed.
  Interventions: Procedure: Ultrasound; Drug: Magnetic Resonance Imaging with Contrast; Procedure: Magnetic Resonance Imaging without Contrast

INTERVENTIONS:
Procedure: Ultrasound — Ultrasounds to be performed on children with central venous catheters
  Other Names: US
Drug: Magnetic Resonance Imaging with Contrast — Contrast-enhanced Magnetic Resonance Imaging (MRI) to be performed on children with central venous catheters
  Other Names: MRI with contrast
Procedure: Magnetic Resonance Imaging without Contrast — Magnetic Resonance Imaging (MRI) to be performed on children with central venous catheters
  Other Names: MRI

SUMMARY:
This protocol will serve as a pilot study to determine the validity and feasibility of contrast enhanced magnetic resonance imaging (MRI) without and with contrast and/or ultrasound (US) for detection of catheter related deep vein thrombosis (DVT) in children

ELIGIBILITY:
Inclusion Criteria:

* Functioning central venous catheter in the upper or lower venous system
* Cohort A: Asymptomatic patients having placement of a new central venous catheter in the last 40±20 days
* Cohort B: Subjects who have experienced symptoms for a CVC-related DVT with a CVC in place or subjects who have been incidentally identified by radiographic imaging (imaging modalities to diagnose an incidental CVC-related DVT may include, but is not exclusive of Echocardiogram, CT scan, MRI, or Ultrasound) performed for other clinical reasons, as having a CVC-related DVT in the veins where the current catheter is placed
* Males and females from full-term newborns to < 18 years

Exclusion Criteria:

* For Cohort A subjects only, present therapeutic dosing of a systematic anticoagulant, systemic thromboprophylaxis or antiplatelet therapy. Local thromboprophylaxis [flushes, low dose infusions of heparin of up to 5 u/kg/hr or locks with heparin, urokinase, t-plasminogen activator] according to standard-of-care at the respective center will be allowed
* Patients unable to undergo contrast enhanced magnetic resonance imaging
* Renal function < 50% of normal for age and size

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (10):
  - Arkansas Children'S Hospital, Little Rock, Arkansas
  - University Of Colorado Denver, Aurora, Colorado
  - Children'S Mercy Hospital And Clinics, Kansas City, Missouri
  - Akron Children'S Hospital, Akron, Ohio
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - The Children'S Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Children'S Hopsital Of Pittsburgh Of Upmc, Pittsburgh, Pennsylvania
  - Dodson Specialty Clinics, Fort Worth, Texas
  - Texas Children'S Hospital, Houston, Texas
  - Ut Health/Gulf States Hemophilia & Thrombophilia Ctr., Houston, Texas
- Local Institution, Buenos Aires, Buenos Aires, Argentina
- Local Institution, Vienna, Austria
- Local Institution, São Paulo, São Paulo, Brazil
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
- Germany (2):
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hanover
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Col. Secc Xvi Tlalpan, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Local Institution, Amsterdam, Netherlands
- Local Institution, Glasgow, Lanarkshire, United Kingdom

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated: 28 February 2011; Study Completed: 10 May 2013. Patients with central venous catheter (CVC) in-place or planned were enrolled. The Study was diagnostic for venous thromboembolism (VTE) and was non-therapeutic.
Pre-assignment Details: 151 participants enrolled; 134 had at least one study-related diagnostic imaging procedure completed or partially completed; 17 enrolled but not identified to a cohort and no study-related imaging procedures performed: Adverse event (2), withdrew consent (1), lost to follow up (1), poor/non-compliance (1), no longer met criteria (3), other (9).
Groups:
- Cohort A: Cohort A included pediatric participants (full-term newborns to <18 years) in which a CVC was recently placed and who were asymptomatic for CVC-related deep vein thrombosis (DVT). Imaging procedures occurred on Day 40 ± 20 days relative to catheter placement (Day 0) and included: ultrasound (US) and magnetic resonance imaging (MRI), with and without contrast enhancement. The MRI and US were to be done within 48 hours of each other. An approved gadolinium contrast agent at a dose which was considered 'state-of-the-art' or standard institutional practice at the specific site and in accordance with the country-specific regulatory guidance was to be used for MRI with contrast. No sedation or anesthesia was to be allowed. Participants who developed symptoms of VTE prior to imaging should have been switched to Cohort B.
- Cohort B: Cohort B included pediatric participants (full-term newborns to <18 years) with a CVC and who were either symptomatic for a CVC-related DVT or had an incidental diagnosis of CVC-related DVT based on radiographic imaging performed for other clinical reasons. Diagnostic imaging procedures, US and MRI (with and without gadolinium contrast enhancement) were to be done within 48 hours of each other or, for those with therapeutic anticoagulation, within 24 hours. Aesthesia/sedation allowed as routine standard of care for participants only if symptomatic for a CVC-related DVT. For those participants symptomatic for a CVC-related DVT, MRI and US were to be initiated within 7 days of symptoms. In those participants with an incidental diagnosis of a CVC-related DVT made by radiographic imaging performed for clinical reasons, MRI and US were to be done within 7 days of the diagnosis of the CVC-related DVT.
- Sub-Study Cohort C: A Sub-study with additional cohort C was initiated to collect diagnostic imaging procedures for the detection of CVC-related DVT in a population < 18 years of age who had a CVC in place and who were scheduled to undergo a contrast enhanced MRI in any part of their body as part of their clinical care and who allowed the diagnostic imaging procedure to include the area around the CVC. Participants who developed symptoms of VTE prior to imaging should have been switched to Cohort B.
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Sub-Study Cohort C
Started | 77 | 14 | 43
Completed | 61 (Completed defined as having completed all 3 study-related imaging procedures.) | 12 (Completed defined as having completed all 3 study-related imaging procedures.) | 37 (Completed defined as having completed all 3 study-related imaging procedures.)
Not Completed | 16 | 2 | 6
Not completed — Participant requested to Discontinue | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other | 12 | 2 | 6

BASELINE CHARACTERISTICS:
Population: All participants who completed or partially completed at least one study-related radiographic procedure.
Groups:
- All Imaged Participants: Baseline parameters for all participants in Cohorts A, B, and C: Pediatric participants (full-term newborns to <18 years) in which a CVC was to be placed or who had a CVC in place. Participants were either asymptomatic (cohort A) or symptomatic for CVC-related deep vein thrombosis (DVT) or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons (cohort B) or participants with a CVC in place and having an MRI with contrast for clinical reasons (Sub-study, cohort C).
Arm/Group | All Imaged Participants
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (4.89)
Age, Customized [Number; unit: participants]
  Less than (<) 2 years | 7
  Between 2 years and <12 years | 64
  Between 12 years and <18 years | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 78
Race/Ethnicity, Customized [Number; unit: participants]
  White | 117
  Black/African American | 7
  Asian | 3
  American Indian or Alaska native | 3
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Who Completed the Study-Related Ultrasound (US) and Magnetic Resonance Imaging (MRI) With and Without Contrast
Description: One set of 3 diagnostic imaging procedures (US, MRI with contrast, and MRI without contrast) was performed for all cohorts. Imaging was performed on Visit 1, which in Cohort A was Day 40 ± 20 days from Day 0, the placement of the central venous catheter (CVC), or if possible within 72 hours after a CVC was removed or lost; Visit 1 in Cohort B was within 7 days of initiation of symptoms of a CVC-related deep vein thromboembolism (DVT) or within 7 days of an incidental diagnosis of CVC-related DVT by radiographic imaging. Cohort C participants had an ultrasound done within 48 hours of the performance of the MRI, which was scheduled for a clinical reason. Note: participants completing each MRI procedure (with contrast or without contrast) could be different participants.
Time Frame: Either Day 40±20 days following the placement of CVC (cohort A) or within 7 days of: symptoms of DVT or incidental diagnosis of CVC-related DVT(cohort B) or Day of MRI + 48 hours (cohort C).
Population: The imaged population included all enrolled participants who had at least 1 study-related diagnostic imaging procedure.
Measure: Number; unit: participants
Groups:
- All Imaged Participants: All participants in Cohorts A, B, and C who had at least 1 radiographic procedure: Pediatric participants (full-term newborns to <18 years) in which a CVC was to be placed or who had a CVC in place. Participants were either asymptomatic (cohort A) or symptomatic for CVC-related deep vein thrombosis (DVT) or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons (cohort B) or participants with a CVC in place and having an MRI with contrast for clinical reasons (Sub-study, cohort C).
Arm/Group | All Imaged Participants
Number analyzed (Participants) | 134
participants
  Completed Ultrasound | 133
  Completed the MRI with Contrast | 113
  Completed the MRI without Contrast | 113
  Completed All 3 Imaging Procedures | 110

2. Primary Outcome: Number of Participants Who Completed the Study-Related Ultrasound and Magnetic Resonance Imaging (MRI) With and Without Contrast, by Cohort and Age Group
Description: Imaging was performed on Visit 1 which was defined for Cohort A as: Day 40 ± 20 days from Day 0, the placement of the central venous catheter (CVC), or if possible within 72 hours after a CVC was removed or lost; Visit 1 defined for Cohort B: within 7 days of initiation of symptoms of a CVC-related deep vein thromboembolism (DVT) or within 7 days of an incidental diagnosis of CVC-related DVT by radiographic imaging. Cohort C participants had an ultrasound done within 48 hours of the performance of the MRI. All 3 imaging procedures, ultrasound, MRI with contrast, MRI without contrast were to be performed on all participants, regardless of the cohort.
Time Frame: as for outcome 1
Population: The imaged population included all enrolled participants who had at least 1 study-related diagnostic imaging procedure.
Measure: Number; unit: participants
Groups:
- Cohort A Newborn to <2Years; Cohort A 2Years to <12Years; Cohort A 12Years to <18Years: Pediatric participants in which a CVC was to be placed (intended stay for 40 ± 20 days) and who were asymptomatic for CVC-related deep vein thrombosis (DVT) were included in Cohort A. Diagnostic imaging procedures: ultrasound (US) and magnetic resonance imaging (MRI), with and without contrast enhancement. The MRI and US were to be done within 48 hours of each other. An approved gadolinium contrast agent at a dose which was considered 'state-of-the-art' or standard institutional practice at the specific site and in accordance with the country-specific regulatory guidance was to be used. No sedation or anesthesia was to be allowed.
- Cohort B Newborn to <2Years; Cohort B 2Years to <12Years; Cohort B 12Years to <18Years: Pediatric participants with a CVC and who were either symptomatic for a CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons were enrolled into Cohort B. Diagnostic imaging procedures, US and MRI, were performed with and without contrast enhancement and were to be done within 48 hours of each other. Aesthesia/sedation allowed as routine standard of care for participants only if symptomatic for a CVC-related DVT. For those participants symptomatic for a CVC-related DVT, MRI and US were to be initiated within 7 days of symptoms. In those participants with an incidental diagnosis of a CVC-related DVT made by radiographic imaging performed for clinical reasons, MRI and US were to be done within 7 days of the diagnosis of the CVC-related DVT. If anticoagulation was started, ultrasound and MRI were to be done within 24 hours of each other.
- Cohort C Newborn to <2Years: Pediatric participants with a CVC in place and having an MRI for clinical reasons were enrolled were enrolled in the substudy, Cohort C. An ultrasound was to be performed around the area of the CVC within 48 hours of the MRI. The MRI was performed both with and without contrast.
- Cohort C 2Years to <12Years; Cohort C 12Years to <18Years: Pediatric participants with a CVC in place and having an MRI for clinical reasons were enrolled in the substudy, Cohort C. An ultrasound was to be performed around the area of the CVC within 48 hours of the MRI. The MRI was performed both with and without contrast.
Arm/Group | Cohort A Newborn to <2Years | Cohort A 2Years to <12Years | Cohort A 12Years to <18Years | Cohort B Newborn to <2Years | Cohort B 2Years to <12Years | Cohort B 12Years to <18Years | Cohort C Newborn to <2Years | Cohort C 2Years to <12Years | Cohort C 12Years to <18Years
Number analyzed (Participants) | 2 | 30 | 45 | 1 | 6 | 7 | 4 | 28 | 11
participants
  Only Ultrasound Completed | 1 | 7 | 6 | 0 | 1 | 0 | 1 | 3 | 0
  Only MRI with contrast Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Only MRI without contrast Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  US and MRI with contrast Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  US and MRI without contrast Completed | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  MRI with and without contrast Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  All 3 Imaging Procedures Completed | 1 | 22 | 38 | 1 | 5 | 6 | 3 | 24 | 10

3. Secondary Outcome: Number of All Participants Identified With Adjudicated DVT Categorized By Presence or Absence of Symptoms at Enrollment
Description: Adjudication was by an ICAC consisting of experienced physicians not involved in the study and blinded to each participant's identity and clinical course. One set of Study-related diagnostic imaging procedures (US, MRI with contrast, and MRI without contrast) was performed for all cohorts. Participants were considered positive for DVT if at least one of the radiographic procedures was positive.
Time Frame: as for outcome 1
Population: All participants who had an adjudicated DVT identified by at lest one study-related radiographic procedure.
Measure: Number; unit: Participants
Arm/Group | All Imaged Participants
Number analyzed (Participants) | 22
Participants
  Symptoms at Enrollment; Adjudicated DVT | 8
  Asymptomatic at Enrollment, Adjudicated DVT | 14

4. Secondary Outcome: Number of Participants With Adjudicated Pulmonary Embolism (PE) Events (Symptomatic or Asymptomatic) Identified During the Study
Description: Signs and symptoms of PE include shortness of breath, pleuritic pain, cough, orthopnea, wheezing, and may have associated signs and symptoms of DVT. In the event a PE was detected while undergoing the study MRI or other imaging procedure required for care of an underlying condition, and the participant did not manifest any signs and/or symptoms of a PE, the event was considered an asymptomatic PE. The participant was managed and further investigated according to the investigator's standard of care. All diagnostic imaging procedures performed, such as contrast-enhanced computer tomography (CT) pulmonary angiogram, nuclear ventilation perfusion lung scan (V/Q scan), were submitted for adjudication as a suspected PE.
Time Frame: Enrollment up to Visit 1 plus 30 days (up to approximately 90 days)
Population: The imaged population included all enrolled participants who had at least one study-related diagnostic imaging procedure.
Measure: Number; unit: participants
Groups:
- Cohort A: Pediatric participants (full-term newborns to <18 years) in which a CVC was to be placed (intended stay for 40 ± 20 days) and who were asymptomatic for CVC-related deep vein thrombosis (DVT) were included in Cohort A. Diagnostic imaging procedures: ultrasound (US) and magnetic resonance imaging (MRI), with and without contrast enhancement. The MRI and US were to be done within 48 hours of each other. An approved gadolinium contrast agent at a dose which was considered 'state-of-the-art' or standard institutional practice at the specific site and in accordance with the country-specific regulatory guidance was to be used. No sedation or anesthesia to be allowed. Participants enrolled in Cohort A and who developed symptoms of a venous thromboembolism (VTE), including a symptomatic DVT or a symptomatic pulmonary embolism (PE) prior to their MRI/US, were switched to Cohort B.
- Cohort B: Pediatric Participants (full-term newborns to <18 years) with a CVC and who were either symptomatic for a CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons were enrolled into Cohort B. Diagnostic imaging procedures, US and MRI, were performed with and without contrast enhancement and were to be done within 48 hours of each other. Aesthesia/sedation allowed as routine standard of care for participants only if symptomatic for a CVC-related DVT. For those participants symptomatic for a CVC-related DVT, MRI and US were to be initiated within 7 days of symptoms. In those participants with an incidental diagnosis of a CVC-related DVT made by radiographic imaging performed for clinical reasons, MRI and US were to be done within 7 days of the diagnosis of the CVC-related DVT. If anticoagulation was started, ultrasound and MRI were to be done within 24 hours of each other.
- Cohort C: Participants with a CVC in place and having an MRI for clinical reasons were enrolled.
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 77 | 14 | 43
participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Required Sedation/Anesthesia With the Study-Related Radiographic Procedures, by Cohort and Age
Description: One set of diagnostic imaging procedures (US and MRI) was to be performed for all cohorts The MRI consisted of MRI venous imaging without contrast enhancement and MRI venous imaging with contrast enhancement.
Time Frame: as for outcome 1
Population: The imaged population included all participants who had at least 1 study-related diagnostic imaging procedure.
Measure: Number; unit: participants
Groups:
- Cohort A Participants <12Years of Age: Cohort A included pediatric participants (full-term newborns to <18 years) in which a CVC was to be placed (intended stay for 40 ± 20 days) and who were asymptomatic for CVC-related deep vein thrombosis (DVT). Diagnostic imaging procedures included: ultrasound (US) and magnetic resonance imaging (MRI), with and without contrast enhancement. The MRI and US were to be done within 48 hours of each other. An approved gadolinium contrast agent at a dose which was considered 'state-of-the-art' or standard institutional practice at the specific site and in accordance with the country-specific regulatory guidance was to be used. No sedation or anesthesia was allowed.
- Cohort A Participants 12Years to 18 Years: Pediatric participants in which a CVC was to be placed (intended stay for 40 ± 20 days) and who were asymptomatic for CVC-related deep vein thrombosis (DVT) were included in Cohort A. Diagnostic imaging procedures: ultrasound (US) and magnetic resonance imaging (MRI), with and without contrast enhancement. The MRI and US were to be done within 48 hours of each other. An approved gadolinium contrast agent at a dose which was considered 'state-of-the-art' or standard institutional practice at the specific site and in accordance with the country-specific regulatory guidance was to be used. No sedation or anesthesia was to be allowed.
- Cohort B Participants <12Years of Age: Cohort B included pediatric participants (full-term newborns to <18 years) with a CVC and who were either symptomatic for a CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons. Diagnostic imaging procedures, US and MRI (with and without contrast enhancement) were to be done within 48 hours of each other. Aesthesia/sedation allowed as routine standard of care for participants only if symptomatic for a CVC-related DVT. For those participants symptomatic for a CVC-related DVT, MRI and US were to be initiated within 7 days of symptoms. In those participants with an incidental diagnosis of a CVC-related DVT made by radiographic imaging performed for clinical reasons, MRI and US were to be done within 7 days of the diagnosis of the CVC-related DVT. If anticoagulation was started, ultrasound and MRI were to be done within 24 hours of each other.
- Cohort B Participants 12Years to 18 Years: Pediatric participants with a CVC and who were either symptomatic for a CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons were enrolled into Cohort B. Diagnostic imaging procedures, US and MRI, were performed with and without contrast enhancement and were to be done within 48 hours of each other. Aesthesia/sedation allowed as routine standard of care for participants only if symptomatic for a CVC-related DVT. For those participants symptomatic for a CVC-related DVT, MRI and US were to be initiated within 7 days of symptoms. In those participants with an incidental diagnosis of a CVC-related DVT made by radiographic imaging performed for clinical reasons, MRI and US were to be done within 7 days of the diagnosis of the CVC-related DVT. If anticoagulation was started, ultrasound and MRI were to be done within 24 hours of each other.
- Cohort C Participants <12Years of Age: A Sub-study with additional cohort C was initiated to collect diagnostic imaging procedures for the detection of CVC related DVT in a population < 18 years of age who had a CVC in place and who were scheduled to undergo a contrast enhanced MRI in any part of their body as part of their clinical care and who allowed the diagnostic imaging procedure to include the area around the CVC.
- Cohort C Participants 12Years to 18 Years: Pediatric participants with a CVC in place and having an MRI for clinical reasons were enrolled in the substudy, Cohort C. An ultrasound was to be performed around the area of the CVC within 48 hours of the MRI. The MRI was performed both with and without contrast.
Arm/Group | Cohort A Participants <12Years of Age | Cohort A Participants 12Years to 18 Years | Cohort B Participants <12Years of Age | Cohort B Participants 12Years to 18 Years | Cohort C Participants <12Years of Age | Cohort C Participants 12Years to 18 Years
Number analyzed (Participants) | 32 | 45 | 7 | 7 | 32 | 11
participants
  Required Sedation for MRI | 0 | 0 | 1 | 0 | 17 | 0
  Required Sedation for US | 0 | 0 | 0 | 0 | 3 | 0

6. Primary Outcome: Number of Participants and Reasons for Non-Completion of Each of the Imaging Procedures, Ultrasound (US), MRI With Contrast and MRI Without Contrast
Description: Bilateral US was attempted but if it could not be completed, a unilateral US was accepted for analysis. Participants who did not complete the MRI procedure with contrast could be different participants from those who did not complete the MRI procedure without contrast. Primary reasons for non-completion of imaging included: technical, investigator decision, child refused, parent refused, child missed appointment, difficulties with anesthesia/sedation, child unable to lie still, problems with contrast administration, and other reasons. Other reasons could include: late to appointment and unable to perform MRI due to time constraints; logistical reasons, parent agreed to only ultrasound at time of consent, schedule delay, equipment not available, difficulty putting patient in correct position. Due to the small numbers of participants in some cohorts, these data were more meaningful with all cohorts grouped together for the total imaged population.
Time Frame: as for outcome 1
Population: Participants had at least 1 radiographic procedure performed but were unable to complete a either an Ultrasound (neither bilateral or unilateral, or could complete only a unilateral US) and/or unable to complete an MRI with contrast and/or unable to complete an MRI without contrast.
Measure: Number; unit: participants
Groups:
- All Imaged Participants: No Ultrasound Performed: Participant had at least one radiographic imaging procedure performed but no study-related US (either bilateral or unilateral) was performed. Pediatric participants in which a CVC was to be placed or who had a CVC in place were included. Participants were either asymptomatic (cohort A) or symptomatic for CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons (cohort B) or participants with a CVC in place and having an MRI with contrast for clinical reasons (Sub-study, cohort C).
- All Imaged Participants: Unilateral Ultrasound Performed: Participant had at least one radiographic imaging procedure performed but a study-related unilateral US instead of a bilateral US was completed. Bilateral US was the protocol-defined procedure but if the participant was not able to complete a bilateral US, then the unilateral US was accepted for evaluation. Pediatric participants in which a CVC was to be placed or who had a CVC in place were included. Participants were either asymptomatic (cohort A) or symptomatic for CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons (cohort B) or participants with a CVC in place and having an MRI with contrast for clinical reasons (Sub-study, cohort C).
- All Imaged Participants: No MRI Without Contrast Performed: Participant had at least one radiographic imaging procedure performed but no study-related MRI without contrast was performed. Pediatric participants in which a CVC was to be placed or who had a CVC in place were included. Participants were either asymptomatic (cohort A) or symptomatic for CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons (cohort B) or participants with a CVC in place and having an MRI with contrast for clinical reasons (Sub-study, cohort C).
- All Imaged Participants: No MRI With Contrast Performed: Participant had at least one radiographic imaging procedure performed but no study-related MRI with contrast was performed. Pediatric participants in which a CVC was to be placed or who had a CVC in place were included. Participants were either asymptomatic (cohort A) or symptomatic for CVC-related DVT or had an incidental diagnosis of CVC-related DVT by radiographic imaging performed for other clinical reasons (cohort B) or participants with a CVC in place and having an MRI with contrast for clinical reasons (Sub-study, cohort C).
Arm/Group | All Imaged Participants: No Ultrasound Performed | All Imaged Participants: Unilateral Ultrasound Performed | All Imaged Participants: No MRI Without Contrast Performed | All Imaged Participants: No MRI With Contrast Performed
Number analyzed (Participants) | 1 | 9 | 21 | 21
participants
  Investigator Decision | 0 | 4 | 2 | 1
  Child Refused Procedure | 0 | 0 | 2 | 3
  Parent Refused Procedure | 0 | 0 | 5 | 5
  Difficulties with Anesthesia/Sedation | 0 | 0 | 3 | 3
  Child Unable to Lie Still | 0 | 0 | 1 | 2
  Problems with Contrast Administration | 0 | 0 | 0 | 1
  Missed Appointment | 1 | 0 | 0 | 0
  Parent or Child Refused to Continue US | 0 | 2 | 0 | 0
  Other reasons | 0 | 3 | 8 | 6

7. Secondary Outcome: Number of Deaths Which Occurred During the Study
Description: Death as an endpoint in a participant with an adjudicated venous thromboembolism (DVT or PE) was summarized, regardless of the cause of the death. The VTE was adjudicated by a blinded central independent adjudication committee.
Time Frame: Enrollment up to last US or MRI plus 30 days (up to approximately 90 days)
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- Cohort A: Pediatric participants (full-term newborns to <18 years) in which a CVC was to be placed (intended stay for 40 ± 20 days) and who were asymptomatic for CVC-related deep vein thrombosis (DVT) were included in Cohort A. Diagnostic imaging procedures: ultrasound (US) and magnetic resonance imaging (MRI), with and without contrast enhancement. The MRI and US were to be done within 48 hours of each other. An approved gadolinium contrast agent at a dose which was considered 'state-of-the-art' or standard institutional practice at the specific site and in accordance with the country-specific regulatory guidance was to be used. No sedation or anesthesia to be allowed. Participants enrolled in Cohort A and who developed symptoms of a venous thromboembolism (VTE), including a symptomatic DVT or a symptomatic pulmonary embolism (PE) prior to their MRI/US, should have been switched to Cohort B.
- Cohort C: A Sub-study with additional cohort C was initiated to collect diagnostic imaging procedures for the detection of CVC-related DVT in a population < 18 years of age who had a CVC in place and who were scheduled to undergo a contrast enhanced MRI in any part of their body as part of their clinical care and who allowed the diagnostic imaging procedure to include the area around the CVC. Participants who developed symptoms of VTE prior to imaging should have been switched to Cohort B.
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 77 | 14 | 43
participants
  Death due to any cause | 0 | 1 | 0
  Death related to study procedures | 0 | 0 | 0

8. Primary Outcome: Number of Participants With an Adjudicated Deep Vein Thrombosis (DVT) Detected By a Study-Related Ultrasound (US) and/or MRI, By Cohort and Age Group
Description: MRI with contrast (c) and without (w/o) contrast (c) enhancement were performed and a US was done within 48 hours of the MRI. Once detected, the DVT was adjudicated and confirmed by an independent central adjudication Committee (ICAC) consisting of experienced physicians not involved in the study and blinded to each participant's identity and clinical course. Participants were considered positive for DVT if at least one of the radiographic procedures was positive. Cohort A: Day 0=day of catheter placement; Day 40 (± 20 days)=day of imaging procedures at Visit 1, or if possible within 72 hours after a CVC is removed or lost. Cohort B Visit 1: within 7 days of initiation of symptoms of a CVC-related DVT (symptoms include but were not limited to: redness, pain/tenderness, swelling, presence of subcutaneous collaterals, catheter occlusion, and the presence of catheter related infection) or within 7 days of an incidental diagnosis of CVC-related DVT by radiographic imaging.
Time Frame: as for outcome 1
Population: The imaged population included all enrolled participants who had at least one study-related diagnostic imaging procedure. n=number of adjudicated images
Measure: Number; unit: participants
Arm/Group | Cohort A Newborn to <2Years | Cohort A 2Years to <12Years | Cohort A 12Years to <18Years | Cohort B Newborn to <2Years | Cohort B 2Years to <12Years | Cohort B 12Years to <18Years | Cohort C Newborn to <2Years | Cohort C 2Years to <12Years | Cohort C 12Years to <18Years
Number analyzed (Participants) | 2 | 30 | 45 | 1 | 6 | 7 | 4 | 28 | 11
participants
  DVTs (n=2,30,45,1,6,7,4,28,11) | 1 | 2 | 4 | 1 | 2 | 5 | 0 | 4 | 3
  Diagnosis by US(n=2,30,45,1,6,7,4,28,11) | 1 | 2 | 4 | 1 | 2 | 4 | 0 | 3 | 2
  Diagnosis by MRI w/o c (n=2,30,45,1,6,7,4,27,11) | 0 | 1 | 2 | 1 | 1 | 3 | 0 | 1 | 1
  Diagnosis by MRI with c (n=2,30,45,1,6,6,4,28,11) | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 2

9. Primary Outcome: All Participants With an Adjudicated Deep Vein Thromboembolism (DVT) By Study-Related Radiographic Procedures That Diagnosed the DVT
Description: Adjudication was by an Independent Central Adjudication Committee (ICAC) consisting of experienced physicians not involved in the study and blinded to each participant's identity and clinical course. One set of 3 study-related diagnostic imaging procedures (US, MRI with contrast, and MRI without contrast) was performed. Participants were considered positive for DVT if at least one of the radiographic procedures was positive.
Time Frame: as for outcome 1
Population: n=participants with an adjudicated DVT identified by a study-related adjudicated radiographic procedure.
Measure: Number; unit: participants
Arm/Group | All Imaged Participants
Number analyzed (Participants) | 22
participants
  Ultrasound (n=22) | 19
  MRI with Contrast (n=20) | 9
  MRI without Contrast (n=21) | 10

ADVERSE EVENTS:
Time Frame: Either Day 40±20 days following the placement of CVC (cohort A) or within 7 days of: symptoms of DVT or incidental diagnosis of CVC-related DVT(cohort B) or Day of MRI + 48 hours (cohort C).
Description: Study initiated February 2011 and Last Patient, Last Visit was May 2013.
Arm/Group | All Imaged Participants
Serious Adverse Events (participants affected / at risk) | 25/134
Other Adverse Events (participants affected / at risk) | 15/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Imaged Participants (N=134)
Device deployment issue (General disorders) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Thrombosis (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Medical device complication (General disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Extravasation (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 1
Skin infection (Infections and infestations) | 1
Asthenia (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Embolism (Vascular disorders) | 1
General physical health deterioration (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Trichosporon infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Thrombosis in device (General disorders) | 3
Venous occlusion (Vascular disorders) | 1
Platelet count decreased (Investigations) | 1
Proctalgia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Imaged Participants (N=134)
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.